CLINICAL TRIAL: NCT03162770
Title: Physiological and Psychological Impact of Mindfulness Meditation Practice on Chronic Hemodialysis Patients
Brief Title: Mindfulness Meditation Practice During Hemodialysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 56794716.1.0000.0071
Record Dates: First submitted 2017-05-03; First posted 2017-05-22 (Actual); Last update posted 2017-05-22 (Actual); Status verified 2017-01

CONDITIONS: Emotional Stress; Hemodialysis Complication
Keywords: mindfulness meditation; hemodialysis; quality of life; stress
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Intervention Model Description: Behavioral: Mindfulness meditation practice This intervention is based on relaxation, well-being promotion, meditation practices and positive psychology principles. The program is being evaluated in hemodialysis session. It will last for 12 weeks, with trainings of 15 to 25 minutes, three times a week.
  No Intervention: Control App This group will observe their psychological and physical condition (levels of stress and well-being) during their daily activities and social interactions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): This group will receive the Mindfulness meditation practice and after that patients will not receive any other intervention.
  Interventions: Behavioral: Mindfulness meditation practice
- No Control Group (No Intervention): Initially this control group will wait and after 12 weeks this group will receive the intervention

INTERVENTIONS:
Behavioral: Mindfulness meditation practice — This intervention is based on relaxation, well-being promotion, meditation practices and positive psychological principles. The program has been conducted during hemodialysis session. It will last for 12 weeks, with duration of 15 to 25 minutes, three times a week.
  Arms: Intervention Group

SUMMARY:
This protocol of meditation is based on mindfulness program proposes to train meditation during the hemodialysis session. The investigators hypothesize that this program offered during hemodialysis session may promote well-being, reduce symptoms of stress and depression reported by the patients, which ultimately may improve biochemical parameters resulting from better adherence to treatment. Objectives: To evaluate the effects of mindfulness meditation practice in patients on chronic hemodialysis, in order to verify if this training can improve symptoms of depression, stress, quality of life and sleep disturbances. Methods: fifty patients will be separated in two groups, twenty five each group, half of them in the control group (CG) and the other half to the intervention group (IG). The patients will be evaluated pre- and pos-protocol.

DETAILED DESCRIPTION:
Introduction: Chronic kidney disease (CKD) affects thousands of people in the world, regardless of gender, race and age. CKD requires dialysis or renal transplant. In the case of dialysis, cardiovascular and infectious events adversely impact the survival and quality of life despite technological advances. Recently, brain-renal interaction has emerged as a key aspect for understanding the neurological disorders-related to CKD, such as cerebrovascular diseases, cognitive impairment, and autonomic, sensory and motor neuropathies. In addition, patients on chronic hemodialysis develop sleep disorders, like insomnia and central apnea, restless leg syndrome, depression, anxiety and stress. Mindfulness meditation practice has been reported to positively affect cardiovascular parameters, since that practice contributes to the decrease in blood pressure levels and premature heart beats occurrence through sympathetic nerve modulation, which collectively may lead to improve the quality of life. Objectives: To evaluate the effects of mindfulness meditation practice in patients on chronic hemodialysis, in order to verify if this training can improve symptoms of depression, stress, quality of life and sleep quality. Methods: fifty patients will be separated in two groups, twenty five each group, half of them in the control group (CG) and the other half in the intervention group (IG). The IG will be enrolled in the meditation protocol, for 12 weeks, 3 days a week during the hemodialysis session, while the CG will wait. Then after the evaluations, the CG will receive the intervention of meditation, while the IG will not receive any intervention. The groups will be evaluate before, 3-and 6-month follow-up periods. We will apply the following instruments: ICED (Index of coexistent diseases), KDQOL (Kidney Disease Quality of Life), BDI (Beck Depression Inventory), PSQI (Pittsburgh Sleep Quality Index), PSS (Perceived Stress Scale), MAAS (Mindful Attention Awareness Scale) and SCS (Self-Compassion Scale).

ELIGIBILITY:
Inclusion Criteria:

* Be a patient at Einstein Dialysis Center
* Have signed the informed consent

Exclusion Criteria:

* Have not signed the informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-03-01 (Estimated); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
Improvement of symptoms of depression, stress, quality of life, sleep disorders, biochemical parameters resulting from better adherence to treatment | up to 12 months
  MAAS (Mindful Attention Awareness Scale):
  Self-report instrument that aims to measure individual differences in the frequency of states of consciousness and mind through time. The greater the more traces of attention (score 15-90).
Improvement of symptoms of quality of life | up to 12 months
  KDQOL (Kidney Disease Quality of Life): Evaluates the perception of quality of life related to renal disease. The closer to 100 the better the perception of quality of life (Score 0-100 on each item- 24 items)
Improvement of symptoms of depression | up to 12 months
  BDI (Beck Depression Inventory):
  From 10 to 18 = mild to moderate depression; From 19 to 29 = moderate to severe depression; From 30 to 63 = severe depression
Improvement of symptoms of sleep disorders | up to 12 months
  PSQI (Pittsburgh Sleep Quality Index):
  Provides a measure of standardized sleep quality, the higher the score, the worse the quality of sleep, PSQI> 5 indicates that the individual is experiencing major difficulties in at least 2 components, or moderate difficulties in more than 3 components
Improvement of symptoms of stress | up to 12 months
  PSS (Perceived Stress Scale):
  Evaluates perceived stress, the greater the more perceived stress (score 0-40).
Improve symptoms of depression and stress | up to 12 months
  SCS (Self-Compassion Scale):
  The answers are given on a likert scale (1- "almost never" to 5 "almost always"), when the answers are not compassionate they must be calculated inversely.
  The scale is subdivided into 6 sub-scales of each of the three mechanisms in their positive and negative characteristics (mindfulness vs. over-identification, self-kindness versus self-judgment, and common humanity vs. isolation). "Global self-pity scores were calculated by inversely encoding the items of self-judgment, isolation, and over-identification, adding up to the six sub-scales.
Assessment of comorbidities | up to 12 months
  ICED (Index of coexistent diseases): The utilization of ICED enables stratifying the dialysis patients according to severity of their comorbidities and it is useful to identify the patients with a greater risk of death and hospitalization, as well as to aid in the forecast of and optimization of resources necessary for their treatment. The ICED aggregates the presence and severity of 19 medical conditions and 11 physical impairments within two scales: the Index of Disease Severity (IDS) and the Index of Physical Impairment (IPI). The final ICED score is determined by an algorithm combining the peak scores for the IDS and IPI. The range of the ICED is from 0 to 3, reflecting increasing severity ( 0 - normal, 1 - mild, 2- moderate, 3- severe).

CONTACTS AND LOCATIONS:
Locations (1):
- Erika Bevilaqua Rangel, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Regular notification when treatment is discontinued, e.g., transplant treatment, death or transfer of dialysis unit